CLINICAL TRIAL: NCT05581550
Title: Somatostatin Receptor Imaging in Nasopharyngeal Cancer, Epstein-Barr Virus (EBV) Related Cancers and Other Rare Tumors
Brief Title: Somatostatin Receptor Imaging in NPC, EBV Related Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: National Cancer Centre Research Fund (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NPC EBV SSTR
Record Dates: First submitted 2021-12-09; First posted 2022-10-14 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Nasopharyngeal Cancer; Epstein-Barr Virus Related Carcinoma
Keywords: Somatostatin; EBV; NPC; Rare Cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET imaging (Other)
  Interventions: Radiation: FDG-PET; Radiation: Galium-68 DOTATATE

INTERVENTIONS:
Radiation: FDG-PET — Patients will be fasted for 6 hours prior to intravenous injection of 370MBq +/- 10% (18)F-fluorodeoxyglucose. Scanning will be performed at an interval of at least 60 minutes following the injection.
Radiation: Galium-68 DOTATATE — 200MBq +/- 10% Galium-68 DOTATATE will be injected intravenously. Scanning will be performed approximately 60 minutes after the injection.

SUMMARY:
The study aims to describe the avidity of somatostatin receptors in locally advanced, metastatic and locally recurrent nasopharyngeal cancer (NPC) and to determine the proportion of NPC patients with high somatostatin receptor density that may benefit from future somatostatin targeted therapeutic trial plans. The investigators also aim to determine the presence of somatostatin receptors in other EBV related cancers.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced, metastatic or locally recurrent NPC that are going for FDG PET as part of their investigations
* Patients that have gone for Ga-68 DOTATATE imaging before are eligible for repeat imaging
* Histologically confirmed NPC
* Above 21 years of age

Exclusion Criteria:

* Patients below 21 years of age
* Pregnant and breast feeding ladies

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Amount of tracer uptake in the tumour lesions of NPC patients | From time of tracer injection to time the scan is performed
  The maximum standardized uptake values (SUVmax) will be measured. If the average SUVmax of all the lesions is more than 10, the patient will be considered to have an overall high somatostatin receptor density.

SECONDARY OUTCOMES:
Amount of tracer uptake in the tumour lesions of patients with EBV related cancers | From time of tracer injection to time the scan is performed
  The maximum standardized uptake values (SUVmax) will be measured. If the average SUVmax of all the lesions is more than 10, the patient will be considered to have an overall high somatostatin receptor density.
Number of somatostatin receptors in patient biopsy samples | Upon signing the informed consent form
Amount of somatostatin circulating tumour cells in patient blood samples | At the time of scan

CONTACTS AND LOCATIONS:
Overall Officials: Wen Long Nei, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore